CLINICAL TRIAL: NCT05079178
Title: Retrospective Clinical Study of the Care and Follow-up in the First Month of Life of Newborns in Level III Services in Alsace From Mothers With COVID-19
Brief Title: Newborns in Level III Services in Alsace From Mothers With COVID-19
Acronym: COVID-Néo
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7863
Record Dates: First submitted 2021-10-14; First posted 2021-10-15 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Newborns of COVID-19 mothers; COVID-19 Pandemic; COVID-19 Virus Disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Very little is known about the impact on the newborn of late pre-partum maternal SARS-CoV-2 infection.

Care without separation of the mother and her newborn with continued breastfeeding has been advocated in France and by the WHO but is being debated in some countries.

Assessment of the development of newborns in their first month of life with this strategy associated with close and secure follow-up.

Importance of reporting the potential benefits / risks of this treatment to guide the care of newborns in a persistent epidemic context in a particularly affected region.

ELIGIBILITY:
Inclusion criteria:

* Newborns born between March 1 and June 30, 2020 to COVID 19
* From positive mothers in Strasbourg University Hospital or Mulhouse Hospital.
* Parents' non-opposition to the analysis of hospitalization data for children contained in the medical file

Exclusion criteria:

- Parents' opposition to the analysis of hospitalization data for children contained in the medical file

Ages: 1 Day to 1 Year | Sex: All
Age Groups: Child
Study Population: Newborns born between March 1 and June 30, 2020 to COVID 19 from positive mothers in Strasbourg University Hospital or Mulhouse Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Retrospective description of the care and follow-up in the first month of life of newborns in level III services in Alsace from mothers with COVID-19 | Files analysed retrospectively from March 01, 2020 to Jun 30, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine et Réanimation du Nouveau-né - Hôpitaux Universitaires de Strasbourg, Strasbourg, France